CLINICAL TRIAL: NCT06843109
Title: Biomarkers as Part of Diagnostic Workup for Alzheimer's Disease: A Feasibility Study in a Canadian Memory Clinic
Brief Title: Biomarkers in a Candian Memory Clinic
Acronym: BioMIND
Status: Enrolling by invitation | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Parkwood Hospital, London, Ontario (Other)
Responsible Party: Sponsor
Other Study IDs: BioMIND
Record Dates: First submitted 2025-01-29; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer's Disease (AD)
Keywords: mild cognitive impairment; dementia; biomarkers
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma will be retained for future research related to biomarkers in Alzheimer's Disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Participants who have not yet completed assessment at Parkwood Institute for memory concerns
- Group B: Participants who have completed assessment at Parkwood Institute for memory concerns.

SUMMARY:
This is a prospective, observational, case control study in a real-world cohort of patients referred by a primary care physician to a tertiary memory clinic for cognitive concerns. This study's main objective is to determine the effect of using standardized criteria (based on eligibility for disease modifying treatment (DMT)) to triage patients towards biological staging of disease with biomarker testing.

ELIGIBILITY:
Inclusion Criteria:

1. Individual with MCI (if not yet diagnosed, individuals with amnestic changes in memory as shown on MoCA)
2. MoCA score must be 18 to 28 inclusive
3. Age 55 to 80 years inclusive
4. Has a study partner that is willing to participate as a source of information and has approximately weekly contact with the subject (contact can be in-person, via telephone or electronic communication). The study partner must have sufficient contact such that the investigator feels the study partner can provide meaningful information about the subject's daily function.
5. Group A - must have a clinical memory assessment appointment scheduled at Parkwood Institute within 18 months of baseline
6. Group B - must have had a clinical memory assessment appointment at Parkwood Institute within 18 months of baseline

Exclusion Criteria:

* 1) Participants who fulfill diagnostic criteria for MCI or dementia/mild or major neurocognitive disorder suspected to be due to any etiology other than AD (eg, MCI/dementia due to frontotemporal lobar degeneration, diffuse Lewy body disease, Parkinson's disease, cerebrovascular disease, normal pressure hydrocephalus, head injury, drug or alcohol abuse/dependence, anoxic brain injury, etc).

  2) Presence of any neurological, psychiatric, or medical conditions associated with a long-term risk of significant cognitive impairment or dementia including, but not limited to, pre-manifest Huntington's disease, multiple sclerosis, Parkinson's disease, Down's syndrome, active alcohol/drug abuse or major psychiatric disorders including, but not limited to, schizophrenia, schizoaffective disorder, or bipolar affective disorder or current episode of major depressive disorder.

  3) Current or history within the past 2 years of psychiatric diagnosis or symptoms (eg, hallucinations, major depression, or delusions) that, in the opinion of the investigator, could interfere with study procedures 4) History of epilepsy, fits, or unexplained blackouts other than vasovagal syncope within 10 years before screening.

  5) Malignant neoplasms within 3 years (except for basal cell or squamous cell carcinoma in situ of the skin) 6) Women of child bearing potential and breastfeeding mothers 7) Individuals who require sedation to complete PET scan. 8) Individuals who are unable to complete assessments in the English language. 9) Individuals who cannot provide consent

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 100 participants will be included from referrals to the Aging Brain and Memory Clinic or Cognitive Neurology. Study investigators will use the CSF and PET scan results to complete the respective surveys. This is a convenience sample so there is not a statistical difference in the number of samples selected as part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of integrating a CSF biomarker into diagnostic decision making for AD. | through study completion, approximately 1 year
  Analysis of resources needed to conduct testing including personnel required, time requirements, space, and resources/equipment

SECONDARY OUTCOMES:
Evaluate the clinical utility of CSF and PET biomarkers in the diagnostic algorithm. | through study completion, approximately one year
  Measured by investigator pre and post biomarker questionnaire indicating clinical suspicion, confidence of clinical suspicion, tests to be ordered, and management plan.
Evaluate the impact of biomarker results on participants | through study completion, approximately one year
  Determined by Participant Pre and Post Biomarker Questionnaire

OTHER OUTCOMES:
Determine the correlation between the plasma biomarker results and CSF results and amyloid PET results | through study completion, approximately one year
  Measured by the percent agreement between plasma biomarker and CSF results and amyloid PET results

CONTACTS AND LOCATIONS:
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will only be available to local site. All study results and conclusions from the study will be shared